CLINICAL TRIAL: NCT07197762
Title: Immunogenicity of a Single Dose of MenB-FHbp or MenACWY-TT/MenB-FHbp in MenB-4C Primed Young Adults
Brief Title: MenB-FHbp or MenACWY-TT/MenB-FHbp Vaccine in MenB-4C Primed Young Adults
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Christina Rostad, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009836; 2025P011916 (Other: Emory IRB)
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neisseria Meningitidis
Keywords: MenACWY-TT/MenB-FHbp [Penbraya, Pfizer]; Meningococcus B; MenB-FHbp [Trumenba, Pfizer]; Neisseria meningitidis serogroup B
MeSH Terms: interventions — MenB-FHbp vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trumenba group (Experimental)
  Interventions: Biological: Trumenba
- Penbraya group (Experimental)
  Interventions: Biological: PENBRAYA

INTERVENTIONS:
Biological: Trumenba — Trumenba is a sterile, recombinant vaccine targeting Neisseria meningitidis serogroup B. It contains two lipidated factor H binding protein (fHbp) variants-A05 from subfamily A and B01 from subfamily B-delivered in a 0.5 mL prefilled syringe. Each dose includes 120 µg of protein (60 µg per variant), 0.018 mg polysorbate 80, and 0.25 mg aluminum as AlPO₄, formulated in histidine-buffered saline at pH 6.0.
  A single intramuscular dose will be administered in the deltoid.
  Arms: Trumenba group
Biological: PENBRAYA — PENBRAYA is a combination vaccine that protects against meningococcal serogroups A, B, C, W, and Y. It consists of two components:
  * A lyophilized MenACWY portion (polysaccharides conjugated to tetanus toxoid)
  * A liquid MenB portion (two recombinant fHbp variants: A05 and B01) Each 0.5 mL dose contains 20 µg of polysaccharides (5 µg per serogroup), 44 µg tetanus toxoid, 120 µg of MenB protein (60 µg per variant), plus stabilizers and aluminum phosphate.
  This will be administered intramuscularly in the deltoid.
  Arms: Penbraya group

SUMMARY:
The goal of this clinical trial is to determine the immunogenicity of certain vaccines in protecting against meningitis B (MenB) in young adults who have previously received a different MenB vaccine.

The main questions it aims to answer are:

* How many participants are protected against four key types of MenB bacteria before and after getting the new vaccine?
* How strong is the immune response after vaccination, and how many people show a noticeable boost in immune response?

DETAILED DESCRIPTION:
Neisseria meningitidis is a human-restricted pathogen that colonizes the nasopharynx and, in rare cases, invades the bloodstream or central nervous system, leading to invasive meningococcal disease (IMD). Clinical manifestations may include meningitis, septicemia, or both. Among the 12 known serogroups, five-A, B, C, W, and Y-account for the majority of global IMD cases. In the United States, serogroups B, C, W, and Y are responsible for approximately 78% of cases across all age groups, with serogroup B being the most prevalent in Europe.

IMD incidence is highest among infants and children under 5 years, adolescents and young adults (particularly ages 16-21), and older adults aged 65 and above.

Vaccination Landscape:

Two monovalent MenB vaccines are currently licensed in the U.S.:

* MenB-4C (Bexsero, GSK)
* MenB-FHbp (Trumenba, Pfizer)

In October 2023, the FDA approved MenACWY-TT/MenB-FHbp (Penbraya, Pfizer), a pentavalent vaccine targeting serogroups A, B, C, W, and Y for individuals aged 10-25 years. The CDC's Advisory Committee on Immunization Practices (ACIP) recommends Penbraya for:

1. Healthy individuals aged 16-23 years when shared clinical decision-making supports MenB vaccination
2. Individuals aged ≥10 years are at increased risk for IMD Due to antigenic differences between MenB-4C and MenB-FHbp (with only one shared antigen), these vaccines are not interchangeable. Continuity with the same manufacturer is required for subsequent doses to ensure immunogenic consistency.

Study Purpose:

This clinical trial aims to characterize the immunogenicity of a single dose of MenB-FHbp (Trumenba) or MenACWY-TT/MenB-FHbp (Penbraya) in young adults previously primed with a two-dose series of the heterologous MenB-4C (Bexsero) vaccine.

The study will evaluate:

Primary Objective: The proportion of participants achieving seroprotection (defined as hSBA titers ≥ lower limit of quantification [LLOQ]) against four MenB indicator strains at baseline and 28 days post-vaccination

Secondary Objectives:

* Geometric mean titers (GMTs) of hSBA responses to the four MenB strains
* Proportion of participants with composite seroprotection (hSBA ≥LLOQ for all four strains)
* Proportion achieving seroresponse (≥4-fold rise in hSBA titers from baseline)

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent before any study procedures are performed.
* Be able to understand and agree to comply with planned study procedures and be available for all study visits.
* Subject is in good health as determined by vital signs, medical history, targeted physical examination (if indicated), and the judgment of the investigator.
* Vaccinated with 2-dose Bexsero primary series at least 2.5 years before vaccination. Must confirm vaccination status and dates of administration through GRITS, healthcare provider, or other official documentation
* Women of childbearing potential must agree to use or have practiced true abstinence2 or use at least one acceptable primary form of contraception from 28 days prior through 28 days after vaccination.
* Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours before vaccination

Exclusion Criteria:

* Subject has an acute illness with fever (temperature ≥100.4 °F) within 72 hours before vaccine administration.
* Subject is currently pregnant or breastfeeding an infant/child.
* Has any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation. (Including acute, subacute, intermittent,t or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial. Chronic medical conditions that are stable, with no escalation in medication doses or new medications administered in the preceding 3 months, will not be considered exclusionary.)
* Presence of self-reported or medically documented significant medical or psychiatric condition(s) as determined by the investigator.
* Received or plans to receive a licensed, live vaccine within 4 weeks before or after the study vaccination.
* Received or plans to receive a licensed, inactivated vaccine within 2 weeks before through 4 weeks after the study vaccination.
* Any previous severe hypersensitivity or anaphylactic reaction to any vaccine or vaccine-related component
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* Received any MenB vaccine within the last 2.5 years before vaccination.
* Received more than 2 doses of Bexsero or any other MenB vaccine(s) (e.g. Trumenba or Penbraya)
* Any known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as participants with congenital or acquired defects in B-cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy >20 mg per day for ≥14 days, or those receiving immunosuppressive therapy. Participants with terminal complement deficiency are excluded from participation in this study.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Any neuroinflammatory condition or autoimmune condition requiring immunomodulatory treatment, including, but not limited to, Guillain-Barré syndrome, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who are seroprotected | Baseline, 28 days post-vaccination
  Percentage of participants who are seroprotected, defined as a human serum bactericidal antibody assay (hSBA) titer ≥LLOQ-Lower limit of quantification (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) for each of the 4 primary MenB indicator strains (A22, A56, B24, and B44) with Trumenba or Penbraya. Serum samples from V1 and V2 will be shipped in batches to Pfizer, where hSBA assays will be performed.

SECONDARY OUTCOMES:
human Serum bactericidal antibody (hSBA) quantity | Baseline, 28 days post-vaccination
  Human serum bactericidal antibody (hSBA) Geometric mean titer will be described for all 4 indicator strains of MenB
Percentage of participants who have composite seroprotection | Baseline, 28 days post-vaccination
  Percentage of participants who have composite seroprotection, defined as achieving an hSBA titer ≥ LLOQ- Lower limit of quantification (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) for all 4 primary MenB test strains combined (composite)
Percentage of participants achieving seroresponse | Baseline to 28 days post-vaccination
  Percentage of participants achieving seroresponse, defined as ≥4-fold rise in hSBA titer

CONTACTS AND LOCATIONS:
Overall Officials: Christina Rostad, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Children's Center-Vaccine Research Clinic, Atlanta, Georgia
  - Hope Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No